CLINICAL TRIAL: NCT07221500
Title: A Single-arm, Phase 2, Open-label, Multicenter Study to Evaluate NX-5948 in Adults With Relapsed/Refractory (R/R) Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) Previously Exposed to a Bruton's Tyrosine Kinase Inhibitor (BTKi) and a B-cell Lymphoma-2 Inhibitor (BCL-2i)
Brief Title: A Study of NX-5948 in Adults With CLL/SLL Previously Treated With a Bruton's Tyrosine Kinase Inhibitor and a B-cell Lymphoma-2 Inhibitor (DAYBreak CLL-201)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nurix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NX-5948-201
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: BTK Degrader; BTK Inhibitor; BCL-2 Inhibitor; B-cell Malignancy; Lymphoma; Bruton's Tyrosine Kinase; NX-5948; Targeted Protein Degradation; Chimeric Targeting Molecule (CTM); Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NX-5948 (Experimental)
  Interventions: Drug: NX-5948

INTERVENTIONS:
Drug: NX-5948 — Oral dose administered once daily. NX-5948 will be given in continuous 28-day cycles.
  Other Names: Bexobrutideg

SUMMARY:
This is a study for patients with relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) who have previously received treatment with a BTK inhibitor (covalent and non-covalent) and a BCL-2 inhibitor. The main purpose of this study is to test if NX-5948 (bexobrutideg) works to treat patients with CLL/SLL. Participation could last up to 5 years, and possibly longer, if the disease does not progress.

DETAILED DESCRIPTION:
The main purpose of this study is to test if NX-5948 works to treat patients with R/R CLL/SLL. NX-5948 is a BTK degrader and works by destroying the BTK protein to stop all its actions. This is different from a BTK inhibitor which works by blocking only the kinase action of BTK. This study aims to answer these questions:

* How well does NX-5948 work to treat patients who have previously received a BTK inhibitor and a BCL-2 inhibitor?
* How safe is NX-5948 and can patients take NX-5948 as long as they need to?
* What is the amount of NX-5948 in the bloodstream over time when given to patients with CLL/SLL?

All patients in the study will receive NX-5948 orally until their cancer gets worse or if there are other reasons to stop taking NX-5948. Patients will have their cancer and other health check-ups regularly while they are taking NX-5948. If a patient's cancer has not gotten worse and they stop taking NX-5948, they will continue to have cancer check-ups until their cancer gets worse.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Confirmed relapsed/refractory CLL/SLL that meets iwCLL criteria for diagnosis and systemic treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Must have received a covalent BTK inhibitor (BTKi), a non-covalent BTKi, and a BCL-2 inhibitor either in separate lines of treatment or in combination
* Measurable disease by radiographic assessment
* Adequate organ and bone marrow function
* Must sign an informed consent form indicating that he or she understands the purpose of the procedures required for the study and is willing to participate

Exclusion Criteria:

* Known or suspected prolymphocytic leukemia or Richter's transformation before entering study
* Investigational agent or anticancer therapy within 5 half-lives or 14 days (whichever is shorter) before planned start of study drug

  * Antibody therapy must stop at least 4 weeks before the first dose of study drug
  * No other systemic anticancer therapy is allowed at the same time as this study; exception: continuation of hormonal therapy for breast and prostate cancer is allowed, if they are not on the list of prohibited concomitant medications in this study
* Radiotherapy within 2 weeks of the first dose of study drug except for focal palliative radiation
* Use of systemic corticosteroids >20 mg/day prednisone or equivalent within the 7 days before start of study drug except for those used as premedication for radio diagnostic contrast
* Use of systemic immunosuppressive drugs other than systemic corticosteroids within 60 days before the first dose of study drug
* Previously treated with a BTK degrader
* Previous chimeric antigen receptor (CAR) T-cell therapy or autologous hematopoietic cell transplant <1 year prior to enrollment
* Thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), stroke, or intracranial hemorrhage within 6 months of planned start of study drug

Note: Other Inclusion/Exclusion criteria may apply as defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate without partial response with lymphocytosis (PR-L) as determined by an Independent Review Committee (IRC) | Up to approximately 5 years
  The percentage of participants with response as determined according to 2018 International Workshop on CLL (iwCLL) guidelines. Response will include complete response (CR)/CR with incomplete marrow recovery (CRi), partial response (PR), and nodular PR.

SECONDARY OUTCOMES:
Objective response rate with PR-L as determined by IRC | Up to approximately 5 years
  The percentage of participants with response as determined according to 2018 iwCLL guidelines. Response will include CR/CRi, PR, and nodular PR.
Objective response rate with and without PR-L as determined by investigator | Up to approximately 5 years
  The percentage of participants with response as determined according to 2018 iwCLL guidelines. Response will include CR/CRi, PR, and nodular PR.
Duration of response as determined by IRC and by investigator | Up to approximately 5 years
  Time from the date of the first response to the date of documented progressive disease or death due to any cause, whichever is earlier
Progression-free survival as determined by IRC and by investigator | Up to approximately 5 years
  Time from the date of the first dose of study drug to the date of documented progressive disease or death due to any cause, whichever is earlier
Complete response rate as determined by IRC and by investigator | Up to approximately 5 years
  The percentage of participants with CR or CRi as determined according to 2018 iwCLL guidelines
Time to response as determined by IRC and by investigator | Up to approximately 5 years
  Time from the start date of study treatment to the date of the first assessment of a response
Overall survival | Up to approximately 5 years
  Time from the start date of study treatment to the date of death from any cause
Number of participants with treatment-emergent adverse events (TEAEs), Grade 3 or higher TEAEs, serious adverse events, and TEAEs leading to study drug discontinuation | Up to approximately 3 years
Number of participants with clinically significant changes from baseline in laboratory parameters | Up to approximately 3 years
  Laboratory parameters may include hematology, clinical chemistry, and urinalysis
Number of participants with clinically significant changes from baseline in vital signs | Up to approximately 3 years
  Vital signs include blood pressure, heart and respiratory rates, pulse oximetry, and temperature
Pharmacokinetic profile of NX-5948 | Up to approximately 1 year
  NX-5948 concentrations in blood samples
Change from baseline in Global Health Status/Quality of Life on the European Organization for Research and Treatment of Cancer QoL Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline and up to approximately 5 years
  Percentage of participants with a clinically meaningful change from baseline using the EORTC QLQ-C30 questionnaire to assess the overall quality of life
Change from baseline in EuroQol-5 Dimensions, 5-level Questionnaire (EQ-5D-5L) | Baseline and up to approximately 5 years
  Percentage of participants with a clinically meaningful change from baseline using the EQ-5D-5L questionnaire to assess health outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Nurix Study Director, Study Director — Nurix Therapeutics, Inc.
Locations (10):
- United States (3):
  - Colorado Blood Institute, Denver, Colorado
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Center South, Austin, Texas
- CHU de Nantes, Nantes, France
- Poland (4):
  - Pratia Hematologia Sp. z o.o., Katowice
  - Pratia S.A., Krakow
  - Aidport Sp. z o.o., Skorzewo
  - Pratia Warszawa / Pratia MTZ, Warsaw
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No